CLINICAL TRIAL: NCT04703192
Title: Single-arm, Phase 2 Study of Valemetostat Tosylate Monotherapy in Subjects With Relapsed/Refractory Peripheral T-Cell Lymphoma (VALENTINE-PTCL01)
Brief Title: Valemetostat Tosylate (DS-3201b), an Enhancer of Zeste Homolog (EZH) 1/2 Dual Inhibitor, for Relapsed/Refractory Peripheral T-Cell Lymphoma (VALENTINE-PTCL01)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-A-U202; 2020-004954-31 (EudraCT Number); jRCT2071200095 (Other: JAPIC)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Peripheral T-Cell Lymphoma; Adult T Cell Leukemia/Lymphoma
Keywords: Relapsed/Refractory Peripheral T-Cell Lymphoma; Adult T-Cell Leukemia/Lymphoma; Valemetostat Tosylate; DS-3201b
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (Experimental): Participants who will receive 200 mg/day valemetostat tosylate and had an eligible peripheral T-cell lymphoma subtype that was confirmed by independent hematopathology central review.
  Interventions: Drug: Valemetostat Tosylate
- Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma (Experimental): Participants who will receive 200 mg/day valemetostat tosylate and had an eligible adult T-cell leukemia/lymphoma subtype that was confirmed by the local pathologist/investigators and by documented positive anti-human T-cell leukemia virus type 1 (HTLV-1) antibody.
  Interventions: Drug: Valemetostat Tosylate

INTERVENTIONS:
Drug: Valemetostat Tosylate — Oral administration of valemetostat tosylate at a dose of 200 mg once daily starting at Cycle 1, Day 1 (continuous for 28-day cycles), until disease progression or unacceptable toxicity
  Other Names: DS-3201b

SUMMARY:
This study will characterize the safety and clinical benefit of valemetostat tosylate in participants with relapsed/refractory peripheral T-cell lymphoma, including relapsed/refractory adult T-cell leukemia/lymphoma.

DETAILED DESCRIPTION:
This study was designed to evaluate the efficacy and safety of valemetostat tosylate monotherapy. The primary objective will evaluate objective response rate of valemetostat tosylate monotherapy as measured by blinded independent central review (BICR) in relapsed/refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Participants ≥18 years of age or the minimum legal adult age (whichever is greater) at the time the informed consent form is signed.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Cohort 1 relapsed/refractory peripheral T-cell lymphoma (PTCL):

  * Diagnosis should be confirmed by the local pathologist; local histological diagnosis will be used for eligibility determination. Participants with the following subtypes of PTCL are eligible according to 2016 WHO classification prior to the initiation of study drug. Any T-cell lymphoid malignancies not listed are excluded. Eligible subtypes include:

    * Enteropathy-associated T-cell lymphoma
    * Monomorphic epitheliotropic intestinal T-cell lymphoma
    * Hepatosplenic T-cell lymphoma
    * Primary cutaneous γδ T-cell lymphoma
    * Primary cutaneous CD8+ aggressive epidermotropic cytotoxic T-cell lymphoma
    * PTCL, not otherwise specified
    * Angioimmunoblastic T-cell lymphoma
    * Follicular T-cell lymphoma
    * Nodal PTCL with T-follicular helper (TFH) phenotype
    * Anaplastic large cell lymphoma, ALK positive
    * Anaplastic large cell lymphoma, ALK negative
* Cohort 2 relapsed/refractory adult T-cell leukemia/lymphoma (ATL) acute, lymphoma, or unfavorable chronic type. Relapsed/refractory ATL should be confirmed by the local pathologist; local diagnosis will be used for eligibility determination. The positivity of anti-human T-cell leukemia virus type 1 (HTLV-1) antibody will be locally determined for eligibility.
* Must have at least one lesion which is measurable in 2 perpendicular dimensions on computed tomography (or magnetic resonance imaging) based on local radiological read
* Documented refractory, relapsed, or progressive disease after at least 1 prior line of systemic therapy.

  * Refractory is defined as:

    * Failure to achieve CR (or CRu for ATL) after first-line therapy
    * Failure to reach at least PR after second-line therapy or beyond
* Must have at least 1 prior line of systemic therapy for PTCL or ATL.

  * Participants must be considered hematopoietic cell transplantation (HCT) ineligible during screening due to disease status (active disease), comorbidities, or other factors; the reason for HCT ineligibility must be clearly documented.
  * In the PTCL cohort, participants with anaplastic large cell lymphoma (ALCL) must have prior brentuximab vedotin treatment.

Exclusion Criteria:

Participants meeting any exclusion criteria for this study will be excluded from this study. Below is a list of the key exclusion criteria:

* Diagnosis of mycosis fungoides, Sézary syndrome and primary cutaneous ALCL, and systemic dissemination of primary cutaneous ALCL
* Diagnosis of precursor T-cell leukemia and lymphoma (T-cell acute lymphoblastic leukemia and T-cell lymphoblastic lymphoma), T-cell prolymphocytic leukemia, or T-cell large granular lymphocytic leukemia
* Prior malignancy active within the previous 2 years except for locally curable cancer that is currently considered as cured, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer.
* Presence of active central nervous system involvement of lymphoma
* History of autologous HCT within 60 days prior to the first dose of study drug
* History of allogeneic HCT within 90 days prior to the first dose of study drug
* Clinically significant graft-versus-host disease (GVHD) or GVHD requiring systemic immunosuppressive prophylaxis or treatment
* Inadequate washout period from prior lymphoma-directed therapy before enrollment, defined as follows:

  * Prior systemic therapy (eg, chemotherapy, immunomodulatory therapy, or monoclonal antibody therapy) within 3 weeks prior or 5 half-lives of the drug, whichever is longer, to the first dose of study drug
  * Had curative radiation therapy or major surgery within 4 weeks or palliative radiation therapy within 2 weeks prior to the first dose of study drug
* Uncontrolled or significant cardiovascular disease, including:

  * Evidence of prolongation of QT/QTc interval (eg, repeated episodes of QT corrected for heart rate using Fridericia's method >450 ms) (average of triplicate determinations)
  * Diagnosed or suspected long QT syndrome or known family history of long QT syndrome
  * History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
  * Uncontrolled arrhythmia (subjects with asymptomatic, controllable atrial fibrillation may be enrolled) or asymptomatic persistent ventricular tachycardia
  * Participant has clinically relevant bradycardia of <50 bpm, unless the participant has a pacemaker
  * History of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers and have no history of fainting or clinically relevant arrhythmia with pacemakers within 6 months prior to Screening
  * Myocardial infarction within 6 months prior to Screening
  * Angioplasty or stent craft implantation within 6 months prior to Screening
  * Uncontrolled angina pectoris within 6 months prior to Screening
  * New York Heart Association Class 3 or 4 congestive heart failure
  * Coronary/peripheral artery bypass graft within 6 months prior to Screening
  * Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg)
  * Complete left bundle branch block
* History of treatment with other EZH inhibitors
* Current use of moderate or strong cytochrome P450 (CYP)3A inducers
* Systemic treatment with corticosteroids (>10 mg daily prednisone equivalents). Note: Short-course systemic corticosteroids (eg, prevention/treatment for transfusion reaction) or use for a non-cancer indication (eg, adrenal replacement) is permissible.
* Known or suspected hypersensitivity to valemetostat tosylate or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2027-02-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (60):
- United States (14):
  - City Of Hope National Medical Center, Duarte, California
  - Stanford University Medical Center - Cancer Clinical Trials Office - ONCOLOGY, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - University Of Colorado Cancer Center, Aurora, Colorado
  - Emory University Hospital - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Memorial Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
- Epworth Healthcare, Richmond, Australia
- Canada (3):
  - BC Cancer - Vancouver Centre, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa
  - University Health Network Princess Margaret Hospital, Toronto
- France (7):
  - CHU de Dijon, Dijon
  - CHRU de Lille - Hôpital Claude Huriez - Maladies du Sang, Lille
  - Centre Lyon Berard - Medical Oncology, Lyon
  - APHP - Hopital Saint Louis, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier Lyon Sud - Hématologie, Pierre-Bénite
  - Institut Universitaire du Cancer de Toulouse-Oncopole (IUCT-Oncopole), Toulouse
- Universitätsklinikum Halle (Saale) - Klinik und Poliklinik für Innere Medizin IV, Halle, Germany
- Italy (5):
  - ASST Papa Giovanni XXIII - Medicina Trasfusionale ed Ematologia - Bergamo, Bergamo
  - A.O.di Bologna Policl.S.Orsola, Bologna
  - PO San Gerardo, ASST Monza, Monza
  - Fondazione Pascale, IRCCS, Istituto Nazionale dei Tumori, Napoli
  - Ospedale S.Maria della Misericordia, AO di Perugia, Università degli Studi di Perugia, Perugia
- Japan (10):
  - National Hospital Organization Nagoya Medical Center - Hematology, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital - Medical Oncology Center, Sapporo, Hokkaido
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - University Hospital - Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Okayama University Hospital, Okayama
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC) (Leiden University Medical Center), Leiden
  - Universiteit Maastricht Academisch Ziekenhuis Maastricht, Maastricht
- South Korea (5):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital - Department of Internal, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center - Hematology-Oncology, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - ICO Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (4):
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital - Hemato-Oncology, Kaohsiung City
  - National Cheng Kung University Hospital - Internal Medicine, Tainan
  - National Taiwan University Hospital - Hematology And Oncology, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Hematology and Oncology - Hematology and Oncology, Taoyuan
- United Kingdom (3):
  - University College London Hospital, London
  - Nottingham City Hospital - Clinical Haematology, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Zinzani PL, Izutsu K, Mehta-Shah N, Barta SK, Ishitsuka K, Cordoba R, Kusumoto S, Bachy E, Cwynarski K, Gritti G, Prica A, Jacobsen E, Feldman T, Guillermin Y, Ennishi D, Yoon DH, Domenech ED, Zain J, Wang J, Kim JS, Poel MV, Jin J, Wu S, Chen Y, Moriyama T, Inoue A, Nakajima K, Horwitz SM. Valemetostat for patients with relapsed or refractory peripheral T-cell lymphoma (VALENTINE-PTCL01): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2024 Dec;25(12):1602-1613. doi: 10.1016/S1470-2045(24)00503-5. Epub 2024 Oct 29. PMID 39486433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 155 participants who met all inclusion criteria and no exclusion criteria were enrolled to receive valemetostat tosylate treatment in 70 study sites in North America, Europe, Asia, and Oceania.
Groups:
- Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL): Participants were administered valemetostat tosylate at a dose of 200 mg/day and had an eligible peripheral T-cell lymphoma .
- Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma (ATCL): Participants were administered valemetostat tosylate at a dose of 200 mg/day and had an eligible adult T-cell leukemia/lymphoma.
Period: Overall Study
Arm/Group | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma (ATCL)
Started | 133 | 22
Completed (Completed = Participants with Ongoing Treatment. Not Completed = Participants who Discontinued Treatment) | 32 | 2
Not Completed | 101 | 20
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 3 | 1
Not completed — Adverse Event | 13 | 2
Not completed — Progressive or Relapsed Disease | 46 | 7
Not completed — Clinical Progression | 19 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Hematopoietic Cell Transplantation | 12 | 1
Not completed — Other | 5 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug. Subjects were analyzed for each cohort.
Groups:
- Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma: Participants were administered valemetostat tosylate at a dose of 200 mg/day and had an eligible adult T-cell leukemia/lymphoma.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma | Total
Number analyzed (Participants) | 133 | 22 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 10 | 63
  >=65 years | 80 | 12 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (12.51) | 62.6 (13.11) | 65.2 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 7 | 49
  Male | 91 | 15 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 34 | 8 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 80 | 1 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response As Assessed by Blinded Independent Central Review After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Description: For the relapsed/refractory peripheral T-cell lymphoma (PTCL) cohort, objective response rate (ORR) is defined as the proportion of participants with a best overall response (BOR) of complete response (CR) or partial response (PR), assessed by blinded independent central review (BICR), among participants with centrally confirmed PTCL eligible histology.
Time Frame: From baseline until disease progression or death (whichever occurs first), up to approximately 23 months
Population: Efficacy Analysis Set for Cohort 1 is defined as all subjects who received at least 1 dose of valemetostat tosylate and had an eligible PTCL subtype that was confirmed by central hematopathology review.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL)
Number analyzed (Participants) | 119
percentage of participants | 43.7 [34.6 to 53.1]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events After Administration of Valemetostat Tosylate Monotherapy (Cohort 2)
Description: Treatment-emergent adverse events (TEAEs) were defined as new AEs or pre-existing conditions that worsen in National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade after the first dose of study drug and up to 30 days after the last dose of study drug.
Time Frame: From the time the informed consent form is signed up to 30 days after last dose, up to 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma
Number analyzed (Participants) | 22
Participants | 22

3. Secondary Outcome: Plasma Concentrations of DS-3201a and CALZ-1809a After Administration of Valemetostat Tosylate Monotherapy
Description: Total and unbound DS-3201a (free form of valemetostat tosylate) and total CALZ-1809a (major metabolite) concentration in plasma will be assessed.
Time Frame: Cycle 1 Day 1, 8, 15 Predose; Cycle 1 Day 1 (1, 2, 4, 5 hours Postdose); Cycle 2 Day 1 Predose; Cycle 3 Day 1 to Cycle 5 Day 1 Predose (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2028-02

4. Secondary Outcome: Duration of Response After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Description: Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of disease progression (progressive or relapsed disease) based on BICR assessments or to death due to any cause, whichever occurs first.
Time Frame: Time from the date of first documented response (CR or PR) until documented disease progression (progressive or relapsed disease) based on BICR assessments or death from any cause (whichever occurs first), up to approximately 56 months
Reporting Status: Not Posted, anticipated posting 2028-02

5. Secondary Outcome: Percentage of Participants With Complete Response After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Description: Complete response rate is the percentage of participants achieving CR as the BOR based on BICR assessments.
Time Frame: From baseline to date of first documented objective response of CR, up to approximately 56 months
Reporting Status: Not Posted, anticipated posting 2028-02

6. Secondary Outcome: Duration of Complete Response After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Description: Duration of complete response is defined as the time from the date of the first documentation of CR to the date of the first documentation of disease progression (progressive or relapsed disease) based on BICR assessments or to death due to any cause, whichever occurs first.
Time Frame: Time from the date of first documented CR until documented disease progression (progressive or relapsed disease) based on BICR assessments or death from any cause (whichever occurs first), up to approximately 56 months
Reporting Status: Not Posted, anticipated posting 2028-02

7. Secondary Outcome: Percentage of Participants With Partial Response After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Description: Partial response rate is the percentage of participants achieving PR as the BOR based on BICR assessment.
Time Frame: From baseline to date of first documented objective response of PR, up to approximately 56 months
Reporting Status: Not Posted, anticipated posting 2028-02

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events After Administration of Valemetostat Tosylate Monotherapy (Cohort 1)
Time Frame: From the time the informed consent form is signed up to 30 days after last dose
Reporting Status: Not Posted, anticipated posting 2028-02

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 30 days after last dose of the study drug, up to 24 months
Description: TEAEs were defined as new AEs or pre-existing conditions that worsen in NCI-CTCAE grade after the first dose of study drug and up to 30 days after the last dose of study drug.
Arm/Group | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma
All-Cause Mortality (participants affected / at risk) | 52/133 | 16/22
Serious Adverse Events (participants affected / at risk) | 53/133 | 15/22
Other Adverse Events (participants affected / at risk) | 120/133 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) (N=133) | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 7 (7) | 3 (3)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Citrobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (2) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (2)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm papilla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) (N=133) | Cohort 2: Relapsed/Refractory Adult T-cell Leukemia/Lymphoma (N=22)
Anaemia (Blood and lymphatic system disorders) | 47 (139) | 11 (41)
Thrombocytopenia (Blood and lymphatic system disorders) | 35 (104) | 4 (13)
Neutropenia (Blood and lymphatic system disorders) | 18 (60) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 38 (56) | 5 (5)
Nausea (Gastrointestinal disorders) | 23 (28) | 4 (5)
Constipation (Gastrointestinal disorders) | 13 (13) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (13) | 3 (4)
Fatigue (General disorders) | 19 (28) | 2 (2)
Pyrexia (General disorders) | 19 (27) | 3 (3)
Asthenia (General disorders) | 17 (22) | 2 (2)
Oedema peripheral (General disorders) | 16 (18) | 2 (2)
COVID-19 (Infections and infestations) | 27 (33) | 4 (4)
Urinary tract infection (Infections and infestations) | 10 (16) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 31 (117) | 9 (40)
Neutrophil count decreased (Investigations) | 18 (54) | 6 (18)
Aspartate aminotransferase increased (Investigations) | 14 (26) | 3 (5)
Alanine aminotransferase increased (Investigations) | 10 (20) | 3 (7)
Weight decreased (Investigations) | 10 (10) | 1 (2)
Blood bilirubin increased (Investigations) | 9 (17) | 1 (4)
Electrocardiogram QT prolonged (Investigations) | 8 (9) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 7 (19) | 2 (4)
White blood cell count decreased (Investigations) | 7 (25) | 4 (8)
Blood creatinine increased (Investigations) | 4 (6) | 2 (6)
Lymphocyte count decreased (Investigations) | 1 (2) | 2 (7)
Decreased appetite (Metabolism and nutrition disorders) | 19 (24) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12) | 3 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (18) | 3 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (10) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (9) | 3 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (7) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 38 (44) | 5 (6)
Headache (Nervous system disorders) | 7 (12) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (19) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (16) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (17) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (11) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04703192/Prot_SAP_000.pdf